CLINICAL TRIAL: NCT06990061
Title: Radiotherapy for BCG-unresponsive Non-muscle-invasive Carcinoma in Situ (CIS) Bladder Cancer
Brief Title: Radiotherapy for BCG-unresponsive Non-muscle-invasive Carcinoma in Situ (CIS) Bladder Cancer: an Open-label, Single-arm, Multicentre, Phase 2 Study
Acronym: BRACE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 2335-GUCG study
Record Dates: First submitted 2025-05-09; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Non-Muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Radiation therapy
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy will be given in 20 fractions of 2.75 Gy (total dose of 55 Gy) covering the whole bladder over 4 weeks in combination.

SUMMARY:
Standard treatment for patients with high-risk NMIBC (high-grade Ta, CIS, or any T1) consists of intravesical Bacillus Calmette-Guerin (BCG) immunotherapy. However, BCG, even administered optimally, does not provide absolute protection and BCG failure is generally considered recurrence or progression during therapy.

Patients who are BCG-unresponsive have a 20-40% risk for progression to muscle-invasive bladder cancer within 5 years, and a 50% risk of developing metastatic disease. For these patients, radical cystectomy with pelvic lymph node dissection and urinary diversion is the standard of care. However, many patients are unable to undergo radical cystectomy because of poor performance status and co-morbidities or decline to undergo surgery.

Although, several phase II studies have shown promising results, none of the drugs are presently available in Europe. An alternative approach is to investigate a possible role for radiotherapy in good prognosis bladder cancer patients. As there is little existing data in NMIBC, the example of bladder preservation in MIBC will be used for guidance.

We aim to evaluate the use of radiotherapy in patients with high-grade non-muscle-invasive bladder cancer who have BCG failure in a single-arm design as per FDA guidelines for this setting. The primary objective is to demonstrate that complete response to treatment 6 months post radiotherapy is seen in more than 30% of patients with BCG-unresponsive, non-muscle invasive carcinoma in situ bladder cancer, unfit or unwilling to undergo radical cystectomy.

Patients with BCG unresponsive non-muscle-invasive bladder cancer according to the EAU guidelines will be treated 20 fractions of 2.75 Gy over 4 weeks with the use of radiosensitisers as per local guidelines. Cystoscopy and urine cytology assessments will be performed at 3 and 6 months from the start of radiotherapy. If either assessment is positive, bladder biopsies or TURBT are required. At the 6-month timepoint, biopsy or TURBT is mandatory. Disease assessments beyond 6 months will be at the treating urologist's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, BCG-unresponsive, high-risk non-muscle-invasive bladder cancer (according to EAU guidelines [2] (see table 1)) °of predominantly (>50%) urothelial histology who were ineligible for or declined to undergo radical cystectomy.

  * Patients with carcinoma in situ with or without high-grade Ta or T1 are allowed if patients with concomitant Ta and T1 tumors have undergone complete TURBT, defined as per standard of care as a visually complete resection. A second TURBT is recommended but not required for patients with T1 tumor.
  * The most recent cystoscopy or TURBT must have been done within 12 weeks before study enrolment.
  * Eastern Cooperative Oncology Group performance status of 0-2
  * Adequate organ function (at minimum WBC > 4.0 × 109/L; platelets > 100 × 109/L; GFR > 25mL/min)
  * 18 years or older
  * Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 72 hrs prior to the first day of radiation.
  * Patients of childbearing / reproductive potential should use adequate birth control measures during the study treatment period and for at least 4 weeks after the last day of radiation. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods include:
  * Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
  * Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
  * Intrauterine device (IUD)
  * Intrauterine hormone-releasing system (IUS)
  * Bilateral tubal occlusion
  * Vasectomized partner
  * Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
  * Before patient 's enrolment, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Evidence of muscle invasive or metastatic urothelial carcinoma
* Evidence of upper urinary tract carcinoma
* Poor bladder function (IPSS >16)
* Hydronephrosis due to tumour in the presence of T1 disease
* Patients on current systemic therapy for bladder cancer
* Patients who have received pelvic external beam radiotherapy within the previous 5 years
* Any known contraindications or allergies to the use of local standard of care radiosensitiser, if applicable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2028-12-01 (Estimated); Study Completion 2031-09-18 (Estimated)

PRIMARY OUTCOMES:
Complete response: each patient will be assessed for his complete response status at 6 months. | 6 months post radiotherapy
  Complete response is defined as at least one of the following:
  Negative cystoscopy and negative (including atypical) urine cytology Positive cystoscopy with biopsy-proven benign or low-grade NMIBC and negative urine cytology.